CLINICAL TRIAL: NCT04357587
Title: Neoadjuvant Immunotherapy in Rectal Cancer: A Pilot Study Examining the Safety and Feasibility of PD-1 Blockade in the Treatment of dMMR or MSI-H Rectal Cancer
Brief Title: Safety and Feasibility of PD-1 Blockade in the Treatment of dMMR or MSI-H Rectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE1220
Record Dates: First submitted 2020-04-20; First posted 2020-04-22 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Rectal Neoplasms
MeSH Terms: conditions — Rectal Neoplasms | interventions — pembrolizumab; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Pembrolizumab (Experimental): Experimental pembrolizumab and SOC external beam radiation and capecitabine
  Interventions: Drug: Pembrolizumab; Radiation: External beam radiation; Drug: Capecitabine

INTERVENTIONS:
Drug: Pembrolizumab — 200 mg intravenously (IV) on days 1, 22, and 43
Radiation: External beam radiation — Daily fractions of 200 cGy, 5 days a week for the first 5 weeks of the study, excluding weekends
Drug: Capecitabine — 825 mg/m2 orally twice a day on days where radiation therapy is given

SUMMARY:
Colorectal cancer is the third most common cancer worldwide and the second leading cause of cancer mortality in the United States. The current standard of care (SOC) for locally advanced rectal cancer includes neoadjuvant chemotherapy and radiation followed by surgery. However, great variability exists in patient's response to neoadjuvant chemoradiotherapy with only about 20-25% of patients achieving a complete response while other patients achieve a partial or no treatment response. The purpose of this study is to test the investigational agent, Pembrolizumab, in combination with SOC radiation and Capecitabine (or 5-Fluorouacil) in treatment of patients with mismatch repair deficient locally advanced rectal cancer.

DETAILED DESCRIPTION:
This study investigates the safety, tolerability, and feasibility of Pembrolizumab, an immunotherapy agent, in combination with SOC radiation and Capecitabine (or 5-Fluorouacil) in treatment of patients with mismatch repair deficient locally advanced rectal cancer. Pembrolizumab is an investigational (experimental) drug that works by enhancing the functional activity of the target lymphocytes (immune cells) to facilitate tumor regression and ultimately immune rejection. Pembrolizumab in combination with radiation and Capcitabine (or 5-Fluorouacil) is experimental because it is not approved by the Food and Drug Administration (FDA) for this specific indication.

The primary objective of this study is to determine the safety, tolerability and feasibility of neoadjuvant pembrolizumab in combination with capectiabine (or 5-Fluorouracil ) in the treatment of patients with MMR-d locally advanced rectal cancer

The secondary objective of this study is to determine the treatment response in MMR-d rectal cancer patients treated with neoadjuvant chemoradiotherapy and Pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

* Must have confirmed rectal adenocarcinoma Defined as, MRI based clinical stage II (T3-4, N0), stage III (T1-4, N+), or oligometastatic locally advanced stage IV that are candidates for curative surgery
* Tumor location at and/or below the peritoneal reflection on MRI.
* Review and discussion at multidisciplinary tumor board with consensus recommendation for neoadjuvant chemoradiation followed by curative-intent surgery. Documented in EPIC tumor board.
* MMR-deficiency confirmed on immunohistochemistry or MSI status confirmed by PCR.
* ECOG Performance status 0-1
* Life expectancy of ≥ 6 months, in the opinion of and as documented by the treating physician.
* Must have normal organ and marrow function as defined below:

  * Hemoglobin ≥ 8.0 g/dL
  * Leukocytes ≥ 3,000/k/uL
  * Absolute neutrophil count ≥ 1,500/k/uL
  * Platelet count ≥ 100,000/k/uL
  * Total bilirubin ≤ 1.3 x institutional upper limit of normal (ULN)
  * AST (SGOT) ≤ 2.5 x institutional upper limit of normal (ULN)
  * ALT (SGPT) ≤ 2.5 x institutional upper limit of normal (ULN)
* Must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior treatment for rectal cancer or prior radiation for other diagnoses to the expected rectal cancer treatment fields.
* Participants receiving any other investigational agents.
* Unresectable primary tumor or unresectable metastatic disease as determined by imaging.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Pembrolizumab or other agents used in this study.
* Participants with uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection
  * Known history of pneumonitis
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or lactating females.
* Female participants who:

  * Are postmenopausal for at least 1 year before the screening visit, OR
  * Are surgically sterile, OR
  * Agree to practice true abstinence from heterosexual contact or agree to use effective contraception without interruption during the study therapy and 90 days after the last dose
* Male participants who: Are surgically sterile, OR Agree to practice true abstinence from heterosexual contact or agree to use effective contraception without interruption during the study therapy and 90 days after the last dose
* HIV-positive participants on combination antiretroviral therapy, participants with active Hepatitis B or C, active tuberculosis, or administration of live vaccine within 30 days of planned start of study therapy will be excluded.
* Participants with a diagnosis of immunodeficiency, active autoimmune disease (including inflammatory bowel disease) or those receiving immunosuppressive therapy within 7 days (other than Prednisone ≤ 5mg daily) prior to the planned start of study treatment will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-08-06 (Actual); Primary Completion 2023-09-25 (Actual); Study Completion 2023-09-25 (Actual)

PRIMARY OUTCOMES:
Rate of adverse events (AEs) as defined by the Common Terminology Criteria for Adverse Events (CTCAE) v5.0 | 30 days after intervention
  Safety endpoint will be defined by rate of AEs as defined by the CTCAE v5.0
Proportion of participants able to complete planned neoadjuvant treatment protocol | 45 days after intervention
  Tolerability as defined by proportion of participants that are able to complete the planned neoadjuvant treatment protocol
Feasibility as defined by proportion of participants with any delay in planned surgery of more than 30 days | 115 days after intervention
  Feasibility as defined by proportion of participants with any delay in the planned surgery of more than 30 days
Treatment response as measured by AJCC tumor regression grade (TRG) | at time of surgical resection, an average of 10 weeks after radiation
  Treatment response as measured by pathologic assessment of treatment response using the AJCC TRG following surgical resection.
  AJCC TRG grading ranges from 0-3:
  0 (complete response): no viable cancer cells
  1. (near complete response): single cells or rare small groups of cancer cells
  2. (partial response): residual cancer with evident tumor regression but more than single cells or rare small groups of cancer cells
  3. (poor or no response): extensive residual cancer with no evident tumor regression.
Treatment response as measured by MRI tumor regression grade | 4-6 weeks before intervention
  Treatment response as measured by MRI tumor regression grade.
  The MRI tumor regression grade uses the following scale:
  1. No/minimal fibrosis visible (tiny linear scar) and no tumor signal
  2. Dense fibrotic scar (low signal intensity) but no macroscopic tumor signal (indicates no or microscopic tumor)
  3. Fibrosis predominates but obvious measurable areas of tumor signal visible
  4. Tumor signal predominates with little/minimal fibrosis
  5. Tumor signal only: no fibrosis, includes progression of tumor
Treatment response as measured by Carcinoembryonic antigen (CEA) blood test | 4-6 weeks before intervention
  Treatment response as measured by CEA levels

CONTACTS AND LOCATIONS:
Overall Officials: David Liska, MD, Principal Investigator — Cleveland Clinic, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose can request the data for meta-analysis by emailing the corresponding author